CLINICAL TRIAL: NCT02247648
Title: Efficacy of Extended-release, Once Daily Tramadol for Post Operative in Ambulatory Shoulder Arthroscopy
Brief Title: Efficacy of Extended-release, Once Daily Tramadol for Post Operative Analgesia in Shoulder Arthroscopy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: unique Protocol ID
Record Dates: First submitted 2014-09-15; First posted 2014-09-25 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2018-02

CONDITIONS: Pain; Vertigo; Nausea; Pruritus
Keywords: tramadol; shoulder surgery; pain; interscalen block; BUPRENORPHINE/HYDROMORPHONE [VA Drug Interaction]
MeSH Terms: conditions — Pain; Vertigo; Nausea; Pruritus | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (Experimental): treatment: tramadol group
  Interventions: Drug: tramadol
- control (Placebo Comparator): control: placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tramadol — Patients from tramadol group received tramadol 100 mg day one, 100 mg day 2, and 200 mg day 3
  Other Names: tridural
  Arms: treatment
Drug: Placebo — Patients from control group received a "shame" tramadol pill on day one, two, and 3
  Arms: control

SUMMARY:
The investigators hypothesize that the use of tramadol will reduce pain and analgesic consumption after arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
The purpose of the study was to evaluate the efficacy of tramadol long acting for post operative pain in patients who had an arthroscopic shoulder surgery in ambulatory setting in comparison with a placebo. The intensity of pain was evaluated on a visual analog scale as the quantity of hydromorphone taken by patients, and the side effects during the first 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 year old
* arthroscopic shoulder surgery on interscalen block
* able to understand the protocol
* inform consent signed

Exclusion Criteria:

* chronic pain or chronic used of narcotics
* Use of IMAO
* Use of ISRS
* Pulmonary chronic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
quantity of hydromorphone consumed | 3 days
  determination of the quantity of hydromorphone consumed at different laps

SECONDARY OUTCOMES:
evaluation of pain (The intensity of pain was evaluated on a visual analog scale) | 3 days
  evaluation of the pain at different laps

OTHER OUTCOMES:
nausea | 3 days
dizziness | 3 days
pruritus | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis Roy, Doctor, Principal Investigator — Head of the Anesthesia Department
Locations (1):
- Institut de chirurgie spécialisée de Montréal, Montreal, Quebec, Canada